CLINICAL TRIAL: NCT03224338
Title: A Phase II, Multicenter, Single-Arm, Open-Label Clinical Trial to Evaluate the Safety and Efficacy of Triple Therapy With Dolutegravir Plus 2 NRTIs, in Treatment-Naïve HIV-2 Infected Subjects
Brief Title: Dolutegravir Plus 2 NRTIs, in Treatment-Naïve HIV-2 Infected Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Blueclinical, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTG-01-01
Record Dates: First submitted 2017-06-06; First posted 2017-07-21 (Actual); Last update posted 2019-09-03 (Actual); Status verified 2019-08

CONDITIONS: HIV II Infection
MeSH Terms: interventions — dolutegravir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- : Dolutegravir (DTG) (Experimental)
  Interventions: Drug: Dolutegravir 50 mg

INTERVENTIONS:
Drug: Dolutegravir 50 mg — Dolutegravir will be used in combination with 2 nucleoside reverse transcriptase inhibitors (NRTIs). The NRTIs used in combination with DTG will be abacavir (ABC) plus lamivudine (3TC) or tenofovir (TDF) plus emtricitabine (FTC), which is in line with the current standard of care. The combination ABC/3TC/DTG will be preferential except in case of hepatitis B co-infection or in case the subject has a positive HLA-B*5701 allele screening assessment.

SUMMARY:
Multicenter, single-arm, open-label clinical trial to evaluate the efficacy, the safety and the tolerability of 50 mg dolutegravir once daily (q.d.) given in combination with 2 NRTIs backbone in HIV-2 positive, treatment-naïve subjects.

DETAILED DESCRIPTION:
Subjects who fulfill all inclusion criteria and none of the exclusion criteria, after giving informed consent, will be eligible for participation in this study. At the Visit 2 (Day1) subjects will receive the study medication and instructions for its administration. Thereafter, subjects will return to the investigational site at week 4, 12, 24, 36 and 48, for efficacy and safety assessments.

Subjects who meet the virologic failure criteria will return to the investigational site approximately one week later to repeat viral RNA testing (Virologic Failure Confirmation visit). If virologic failure is confirmed and the viral load meets the criteria for resistance testing, viral resistance testing will then be performed.

ELIGIBILITY:
Inclusion Criteria:

* A subject is eligible for the study if he/she fulfills all of the following inclusion criteria:

  1. Able to understand and willing to comply with all the requirements of the study, as confirmed by giving voluntary written informed consent for participation.
  2. Male or female gender.
  3. Age ≥ 18 years on the day of signing the informed consent.
  4. HIV-2 positive as determined by a positive result in the respective assay.
  5. CD4 count ≤500 cells/mm3 (in case of undetectable baseline HIV-2 viral load); and/or classified as B- or C-stage, by the HIV disease staging and classification system of Centers for Disease Control and Prevention (CDC); and/or have detectable viral load irrespective of CD4 count; and/or have other medical conditions / co-morbidities in which treatment is considered, according to European AIDS Clinical Society (EACS) and national guidelines;
  6. Naïve to ART including investigational antiretroviral agents .
  7. Considered clinically stable with no signs or symptoms of active infection, at the time of entry into the study (i.e., clinical status and all chronic medications should be unchanged for at least 2 weeks prior to the start of treatment in this study), in the opinion of the investigator.
  8. If woman or man with reproductive potential, agrees to adopt one of the following effective contraceptive methods throughout the study:

     1. True abstinence, if this is in line with the preferred and usual lifestyle of the subject [Period abstinence (e.g., abstinence only on certain calendar days, abstinence only during ovulation period, use of symptothermal method, use of post-ovulation methods) and withdrawal are not acceptable methods of contraception].
     2. Use of an acceptable method of birth control throughout the study (either by subject or subject's partner). Acceptable methods of birth control are: oral contraceptive, intrauterine device (IUD), diaphragm with spermicide, contraceptive sponge, condom, vasectomy. All forms of hormonal contraception are acceptable. However, the investigator should consult local prescribing information for guidance on the use of hormonal contraceptives with background ART as some antiretrovirals have clinically significant drug interactions with these products.

NOTE: A subject who is not of reproductive potential , is not sexually active, whose current partner(s) is/are not of reproductive potential, or whose sexual activity is exclusively homosexual is eligible without requiring the use of contraception. However, use of barrier methods of contraception is strongly encouraged to reduce the risk of HIV-2 transmission during sexual contact.

Exclusion Criteria:

* A subject is not eligible for the trial if he/she fulfills any of the following exclusion criteria:

  1. History or presence of allergy to the study drugs or their components.
  2. HIV-1 infection or HIV-1/HIV-2 dual infection.
  3. History or current evidence of any condition, therapy, laboratory abnormality or other circumstance that might confound the results of the study, or interfere with the subject's participation for the full duration of the study, such that it is not in the best interest of the subject to participate.
  4. Documented or known resistance to DTG and/or NRTIs.
  5. Treatment with systemic immunosuppressive therapy or immune modulators within 30 days prior to treatment in this study or is anticipated to need them during the course of the study.

     NOTE: "Short courses" of corticosteroids (e.g., as for asthma exacerbation) will be allowed. "Short courses" mean a use of corticosteroids for less than 7 days.
  6. Requiring or is anticipated to require any of the prohibited medications while in the study (dofetilide, inducers of CYP3A4, including phenobarbital, phenytoin, carbamazepine and rifampicin).

     NOTE: Subjects must discontinue phenobarbital, phenytoin, carbamazepine, and rifampicin at least 14 days prior to the treatment phase of the study.
  7. Current (active) diagnosis of tuberculosis.
  8. Alanine aminotransferase (ALT) ≥5 times the upper limit of normal (ULN), or ALT ≥3xULN and bilirubin ≥1.5xULN (with >35% direct bilirubin).
  9. Moderate to severe hepatic impairment (Class B or greater) as determined by Child-Pugh classification .
  10. If subject eligible to receive Tivicay®: Unstable liver disease (as defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice), cirrhosis, known biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
  11. Estimated creatinine clearance <50 mL/min at time of screening, based on Cockcroft-Gault equation .
  12. Current (active) diagnosis of acute hepatitis due to any cause. NOTE: Subjects with chronic hepatitis B and C may enter the study as long as they fulfil all entry criteria, have stable liver function tests, and have no significant impairment of hepatic synthetic function (significant impairment of hepatic synthetic function is defined as a serum albumin <2.8 g/dL in the absence of another explanation for the abnormal laboratory value) at the time of enrollment.
  13. Under treatment for a viral infection other than HIV-2, such as hepatitis B, with an agent that may be active against HIV-2, including but not limited to 3TC, TDF or entecavir, unless the treatment with these agents occurred prior to the diagnosis of HIV.
  14. Anticipated need for Hepatitis C virus (HCV) therapy with interferon and/or ribavirin during the study.
  15. Positive HLA-B*5701 allele screening assessment and is also not eligible for treatment with the other acceptable NRTIs (TDF/FTC).
  16. Significant suicidality risk, according to the investigator's judgment. NOTE: Recent history of suicidal behavior and/or suicidal ideation may be considered as evidence of serious suicide risk.
  17. Participation in a study with an investigational compound/device within 30 days of signing informed consent or anticipates participating in such a study involving an investigational compound/device during the course of this study.
  18. If woman, she is pregnant, breastfeeding, or expecting to conceive at any time during the study.
  19. If woman, she is expecting to donate eggs at any time during the study.
  20. If man, expecting to donate sperm at any time during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Efficacy analysis- treatment efficacy, as measured by the "overall treatment success defined as proportion of patients with "global success" at week 48. | 48 Weeks
  The primary objective of this study is to evaluate the efficacy of DTG in combination with two NRTIs [ABC/3TC or TDF/FTC] in the treatment of HIV-2 treatment-naïve subjects, as measured by the proportion of subjects achieving a plasma viral load of <40 copies/mL and/or by the change from baseline in CD4 cell count and in CD4/CD8 ratio at Week 48. Global success" is a composite variable defined as a plasma HIV-2 RNA viral load <40 copies/mL and a delta of CD4 depending on the initial CD4 count (CD4 delta >+100 cells/mm3 for initial CD4s ≤ 500 cells/mm3; or CD4delta > +50 cells/mm3 for initial CD4s > 500 cells/mm3).

SECONDARY OUTCOMES:
Study treatment immunological effect | 12, 24 and 48 Weeks
  To evaluate the study treatment immunological effect, as measured by the change from baseline in CD4 cell count and the CD4/CD8 ratio at Week 48.
  as measured by the change from baseline in CD4 cell count and the CD4/CD8 ratio at Week 48. Change from Baseline in CD4 Cell Count and CD4/CD8 ratio Change from baseline in CD4 cell count and the CD4/CD8 ratio will be estimated at each time point with CD4 and CD8 cell count collection with a key interest at Week 12, 24 and 48.
Study treatment immunological effect | 12, 24 and 48 Weeks
  Proportions of subjects achieving HIV-2 RNA < 40 copies/mL. The proportions of subjects achieving HIV-2 RNA <40 copies/mL will be estimated at Week 12, 24 and 48.
Safety and tolerability of the study treatment, as assessed by review of the accumulated safety data. | 24 weeks or rebounder at least one week apart afte rinitial response
  The following clinical and laboratory adverse experiences will be summarized:
  Subjects with at least one adverse experience. Subjects with at least one drug related adverse experience. Subjects with at least one serious adverse experience. Subjects with at least one serious and drug related adverse experience, Subjects who discontinued study therapy due to an adverse experience.

OTHER OUTCOMES:
Antiretroviral activity | 48 Weeks
  The exploratory objective of this study is to evaluate the antiretroviral activity of DTG in combination with two NRTIs [ABC/3TC or TDF/FTC] against HIV-2, as measured by the Time to Virologic Response (TVR)
Antiretroviral activity | 48 Weeks
  The exploratory objective of this study is to evaluate the antiretroviral activity of DTG in combination with two NRTIs [ABC/3TC or TDF/FTC] against HIV-2, as measured by the Time to Loss Of Virologic Response (TLOVR).

CONTACTS AND LOCATIONS:
Locations (6):
- Portugal (6):
  - Centro Hospitalar de Lisboa Central Hospital Curry Cabral, Lisbon
  - Centro Hospitalar de Lisboa Ocidental Hospital de Egas Moniz, Lisbon
  - Centro Hospitalar Lisboa Norte Hospital de Santa Maria, Lisbon
  - Hospital Beatriz Ângelo Loures, Lisbon
  - Hospital Garcia de Orta, Lisbon
  - Hospital Professor Doutor Fernando Fonseca Amadora, Lisbon

REFERENCES:
- [Derived] Pacheco P, Marques N, Rodrigues P, Mansinho K, Maltez F, Janeiro N, Franco C, Trigo D, Batista J, Duque L, Lopes MJ, Aleixo MJ, Silva AR, Tavares R, Alves J, Peres S, Povoas D, Lino S, Gomes P, Araujo V, Lopes C. Safety and Efficacy of Triple Therapy With Dolutegravir Plus 2 Nucleoside Reverse Transcriptase Inhibitors in Treatment-Naive Human Immunodeficiency Virus Type 2 Patients: Results From a 48-Week Phase 2 Study. Clin Infect Dis. 2023 Sep 11;77(5):740-748. doi: 10.1093/cid/ciad339. PMID 37288954